CLINICAL TRIAL: NCT00225459
Title: Does Spiritual/Religious Commitment Mediate the Relationship Between Mood Variability and Suicidal Ideation.
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other)
Responsible Party: Principal Investigator, Marilyn Baetz, Professor of Psychiatry, University of Saskatchewan
Other Study IDs: Beh-REB 05-18
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Anxiety Disorder; Mood Disorder
Keywords: Religious psychology; Anxiety disorder; Mood disorder; Suicide
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Suicide

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine whether or not spiritual and/or religious commitment affects mood variability and thoughts of suicide.

First we hypothesize that among patients with depressive symptoms, those who have higher religious/spiritual (R/S) commitment will have less suicidal ideation and less mood variability. Second, we hypothesize that higher mood variability will be associated with more suicidal ideation. Finally, dependent on the first two hypotheses, we propose that R/S commitment will mediate the relationship between mood variability and suicidal ideation.

DETAILED DESCRIPTION:
The suicide rate has not changed dramatically in the recent past, despite advances in psychiatric and mental health treatment, suicide prevention and awareness programs, and reorganization of health services. Depression and the mood disorders which may affect 15% of the population are the conditions most associated with high suicide rates (in addition to psychotic conditions that are relatively rare). Research findings into specific conditions within the depressive disorders that might predict suicidal tendencies are sparse, except for other common comorbid conditions such as panic and alcohol abuse. Research into risks and protective factors has infrequently included religious and spiritual variables that have been associated with decreased rates of depression, suicide, suicide attempts and suicidal ideation.

An inverse relationship between religion and suicide has been found in regional, national, and cross-national studies. Analyzing data from the 1993 Mortality Followback Survey in the US, frequency of religious activities reduced the odds of dying by suicide even after controlling for the frequency of social contact; in 584 deaths by suicide compared with 4279 natural deaths. A Canadian study of 261 Census divisions found the absence of religious affiliation to be an important predictor of death by suicide.

There are no known studies examining mood variability and religion, or spirituality directly. A number of studies however have examined personality attributes and religiosity. The personality style of neuroticism includes moodiness and negative emotionality with the concept of mood reactivity being germane to its construct. Neuroticism is highly correlated with depression and may be a higher order factor in the "internalizing disorders" which include the depressive and anxiety disorders.

The objective of this study is to answer the question "Does R/S mediate the relationship between mood variability and suicidal ideation?" In an effort to achieve that objective, there are three questions that must be answered in this population which in themselves are significant contributions to the research literature.

1. Is there an association between mood variability and suicidal ideation?
2. Is there an association between mood variability and religion?
3. Is there an association between religion and suicidal ideation?

We hypothesize that those who endorses higher religious/spiritual commitment as measured by daily spiritual experiences, positive religious coping, and personal devotion, will have less suicidal ideation, and less mood variability. Secondly, we hypothesize that higher mood variability will be associated with more suicidal ideation. Finally, dependent on the first two hypotheses, we propose that R/S commitment will mediate the relationship between mood variability and suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients.
* DSM-IV defined major depression.
* Comorbid anxiety, bipolar spectrum, and schizoaffective (depressive type).
* Males and females between the ages of 18 and 70.

Exclusion Criteria:

* Involuntary patients.
* In/out patients with current psychosis.
* In/out patients with neurological impairment.
* In/out patients with current substance dependence.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is psychiatric inpatients and outpatients with depressive symptoms between the ages or 18 and 70. Co-morbid anxiety, bipolar spectrum, and eating disorders will be allowed. Involuntary patients and those with psychosis, organic brain impairment, and current substance dependence will be excluded. We will recruit patients prospectively, as they attend psychiatrists' clinics and are admitted to hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2005-06; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Baetz, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan Department of Psychiatry, Saskatoon, Saskatchewan, Canada